CLINICAL TRIAL: NCT03916055
Title: Clinical and Cost-effectiveness of Internet-delivered Behaviour Therapy for Children and Adolescents With Tourette's Disorder: a Single-blind Randomised Controlled Trial
Brief Title: Internet-delivered Behaviour Therapy for Children and Adolescents With Tourette's Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government); Uppsala University (Other)
Responsible Party: Principal Investigator, David Mataix-Cols, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/1788-31/2
Record Dates: First submitted 2019-04-04; First posted 2019-04-16 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Tourette's Disorder; Persistent (Chronic) Motor or Vocal Tic Disorder
Keywords: Tourette syndrome; Tourette; Tics; Behavior therapy; ERP; Internet; Self-help
MeSH Terms: conditions — Tourette Syndrome; Bronchiolitis Obliterans Syndrome; Tic Disorders; Tics

STUDY DESIGN:
Intervention Model Description: Single-blind parallel-group randomised controlled superiority trial.
Who Masked: Outcomes Assessor
Masking Description: Assessors conducting post- and follow-up assessments will be blind to treatment allocation, for the full duration of the trial. At each follow-up assessment, participants will be reminded by their assessor to not reveal their arm allocation. To measure blinding integrity, all assessors will record whether the participating families inadvertently reveal their group allocation, and subsequently guess each participant's treatment allocation at each assessment point, and motivate their choice. If the treatment allocation is accidently revealed, that very part will be cut out of the video recording, and a new blind assessor will watch the video and conduct the assessment that will be used in the trial. Subsequent assessments for that participant will then be conducted by a different assessor (than the first one; blind to treatment allocation), where possible. The blinding will be broken after the trial's final participant has finished her/his 3-month follow-up assessment (primary endpoint).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposure and response prevention (ERP) (Experimental): Therapist-guided and parent-guided internet-delivered exposure and response prevention (ERP)
  Interventions: Behavioral: Exposure and response prevention (ERP)
- Education on tics (Active Comparator): Therapist-guided and parent-guided internet-delivered education on tics
  Interventions: Behavioral: Education on tics

INTERVENTIONS:
Behavioral: Exposure and response prevention (ERP) — The intervention consists of 10 modules/chapters for children/adolescents, delivered over 10. Each of the 10 modules includes age-appropriate texts, animations and exercises. The intervention is primarily based on ERP techniques. During the treatment, participants are instructed to practice suppressing their tics, this is known as 'response prevention'. Then, with the help of their caregiver/parent, the participant is instructed to provoke premonitory urges (a sensation usually felt before a tic is expressed), while still suppressing tics, which is known as 'exposure'.
  The parent is provided with her/his own separate login to the internet platform, which consists of 10 separate modules/chapters. The parent intervention consists mainly of information regarding parent coping strategies, social support and functional analysis relating to tics. Both the child/adolescent and the parent have individual access to the same therapist.
  Other Names: BIP TIC
  Arms: Exposure and response prevention (ERP)
Behavioral: Education on tics — The active comparator is designed to match the experimental intervention in all aspects except for the module content (same platform, same treatment length, same therapist support etc.). The intervention consists mainly of psychoeducational information about TD/PTD and common comorbid conditions, and reviews the definition of tics, natural history, common presentations, prevalence, aetiology, risks and protective factors, strategies for describing tics to other people, among others. Problem-solving and development of expertise in tic disorders is emphasised. The intervention does not include any information on ERP or functional analysis and interventions.
  As in the experimental intervention, the parent is provided with her/his own separate login to the internet platform. The parent intervention consists mainly of information regarding parent coping strategies and social support. Both the child and the parent have individual access to the same therapist.
  Arms: Education on tics

SUMMARY:
The purpose of this trial is to evaluate the clinical efficacy, 12-month durability, and cost-effectiveness of BIP TIC - a therapist-guided and parent-guided internet-delivered behavioural intervention for children and adolescents with Tourette's Disorder and Persistent (Chronic) Motor or Vocal Tic Disorder.

DETAILED DESCRIPTION:
Primary objective: To determine the clinical efficacy of BIP TIC (Andrén et al., 2019; a therapist-guided and parent-guided, internet-delivered behavioural intervention for Tourette's Disorder (TD) and Persistent (Chronic) Motor or Vocal Tic Disorder (PTD), for reducing tic severity (as measured by the primary outcome variable Yale Global Tic Severity Scale [YGTSS] Total Tic Severity Score [TTSS]) in children and adolescents with TD/PTD, compared with a control intervention (therapist-guided and parent-guided internet-delivered education on tics).

Secondary objectives: To establish the 12-month durability of the treatment effects, and to assess the cost-effectiveness of BIP TIC, compared with therapist-guided and parent-guided internet-delivered education on tics, from a societal perspective.

Type of trial: Single-blind parallel-group randomised controlled superiority trial.

Trial design and methods: All potential participants are initially screened via the telephone, or in some cases at the clinic. This is followed by an inclusion assessment conducted either at the clinic or via the videoconference software Zoom. Participants who are eligible and have consented will be randomised into one of two trial arms. In the experimental arm, participants receive 10 weeks of therapist-guided and parent-guided internet-delivered exposure and response prevention (ERP). In the control arm, participants receive 10 weeks of therapist-guided and parent-guided internet-delivered education on tics. Participants will complete outcome measures at baseline, mid-treatment (3 and 5 weeks post-baseline), post-treatment (10-weeks post-baseline) and 3, 6 and 12 months post-treatment. To allow for holidays or periods of sick leave, it is possible to extend the duration of the treatment from 10 to a maximum of 12 weeks (of which only 10 weeks will include therapist support). In these cases, the listed time frames in the "Outcome Measures" section will be extended with the equivalent number of weeks.

The primary outcome variable is the Total Tic Severity Score (TTSS) of the Yale Global Tic Severity Scale (YGTSS), and the primary endpoint is the follow-up 3-months post-treatment. For secondary outcomes, see section below. Follow-up assessments will be conducted at the clinic or via Zoom videoconference software, in both cases complemented with online questionnaires.

Planned trial sites: All assessments and delivery of treatment will be administrated from a single site in Stockholm, the Child and Adolescent Psychiatry Research Center. Several collaborating counties all across Sweden will assist on referring potential participants to the Stockholm site for inclusion in the trial.

Sample: 220 participants.

Statistical methodology and analysis: Data will be analysed using a pre-specified intention-to-treat statistical analysis plan.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 9 to 17 years. Confirmed by the caregiver and subsequently by the patient record system TakeCare.
2. A diagnosis of Tourette's Disorder or Persistent (Chronic) Motor or Vocal Tic Disorder, based on the 5th edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5). Confirmed by the assessor at the face-to-face or videoconference inclusion assessment.
3. A Total Tic Severity Score (TTSS) of >15 (or >10 if only motor or vocal tics, but not both, have been present the last week) on the YGTSS. Confirmed by the assessor at the face-to-face or videoconference inclusion assessment.
4. A minimum of one available caregiver (parent) to support the child/adolescent throughout the treatment. Confirmed by the caregiver at the telephone screening or/and face-to-face or videoconference inclusion assessment.
5. Regular access to a desktop or laptop computer connected to the internet, with the ability to receive e-mails, as well as a mobile phone to receive SMS (one of each is enough per family). Confirmed by the caregiver at the telephone screening or/and face-to-face or videoconference inclusion assessment.

Exclusion Criteria:

1. Previous behaviour therapy for tics, for a minimum of eight sessions with a qualified therapist within the 12 months prior to assessment. Confirmed by the caregiver at the telephone screening or/and face-to-face or videoconference inclusion assessment.
2. Simultaneous psychological treatment for Tourette's Disorder or Persistent (Chronic) Motor or Vocal Tic Disorder. Confirmed by the caregiver at the telephone screening or/and face-to-face or videoconference inclusion assessment.
3. Initiation or adjustment of any psychotropic medication for Tourette's Disorder or Persistent (Chronic) Motor or Vocal Tic Disorder within the eight weeks prior to assessment. Confirmed by the caregiver at the telephone screening or/and face-to-face or videoconference inclusion assessment.
4. A diagnosis of organic brain disorder, intellectual disability, autism spectrum disorder, psychosis, bipolar disorder, anorexia nervosa, or alcohol/substance dependence. Confirmed by the assessor at the telephone screening or/and face-to-face or videoconference inclusion assessment, with help of information from the caregiver and the child/adolescent, and the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID) interview.
5. Immediate risk to self or others, requiring urgent medical attention, such as suicidality, or self-injurious tics. Confirmed by the assessor at the telephone screening or/and face-to-face or videoconference inclusion assessment.
6. Child or caregiver (parent) not able to read and communicate in Swedish. Confirmed by the caregiver or assessor at the telephone screening or/and face-to-face or videoconference inclusion assessment.
7. A participant with a close relationship to the child/adolescent (e.g., sibling, cousin) has already been included in the trial.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 221 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
Yale Global Tic Severity Scale (YGTSS) Total Tic Severity Score (TTSS) | Baseline; week 10; 3-month follow-up; 6-month follow-up; 12-month follow-up.
  Change in tic severity (motor and/or vocal tics) (range 0-50 points) from week 0 (baseline) to week 10 (post-treatment), 3-month follow-up (after post-treatment), 6-month follow-up and 12-month follow-up. The primary endpoint is the 3-month follow-up. The TTSS can also be divided into separate severity scores for motor tics (range 0-25 points) and vocal tics (range 0-25 points). When summed, these two scores comprise the TTSS (range 0-50 points). A higher value represents a greater tic severity. Clinician-rated, semi-structured interview.

SECONDARY OUTCOMES:
Yale Global Tic Severity Scale (YGTSS) Impairment | Baseline; week 10; 3-month follow-up; 6-month follow-up; 12-month follow-up.
  Impairment score (range 0-50 points) of the YGTSS. Used to assess tic specific impairment. Clinician-rated, semi-structured interview.
Clinical Global Impression - Severity (CGI-S) | Baseline; week 10; 3-month follow-up; 6-month follow-up; 12-month follow-up.
  Used to provide an overall rating of the tic disorder severity. Clinician-rated.
Clinical Global Impression - Improvement (CGI-I) | Week 10; 3-month follow-up; 6-month follow-up; 12-month follow-up.
  Used to assess global improvement. Clinician-rated. Treatment response in the trial is operationalised as scores of "very much improved" (1) or "much improved" (2) on the CGI-I.
Children's Global Assessment Scale (CGAS) | Baseline; week 10; 3-month follow-up; 6-month follow-up; 12-month follow-up.
  Used to assess global improvement. Clinician-rated.
internet intervention Patient Adherence Scale (iiPAS) | Mid-treatment (5 weeks post-baseline); week 10.
  Used to assess the child/adolescent's adherence to the internet-delivered treatment. Clinician-rated.
Therapist platform time | Week 10.
  Therapist platform time is automatically logged in the internet treatment platform. Separate data for children and parents.
Therapist telephone time | Week 10.
  Therapist telephone time is manually logged in a spreadsheet throughout the trial. Separate data for children and parents.
Number of completed chapters in the internet treatment platform | Week 10.
  Number of completed chapters is automatically logged in the internet treatment platform. Separate data for children and parents.
Number of logins to the internet treatment platform | Week 10; 12-month follow-up.
  Number of logins is automatically logged in the internet treatment platform. Separate data for children and parents.
Average time between logins to the internet treatment platform | Week 10.
  Average time between logins is automatically logged in the internet treatment platform. Separate data for children and parents.
Average pages visited in the internet treatment platform | Week 10.
  Average pages visited in the internet treatment platform. Separate data for children and parents.
Number of characters submitted in the internet treatment platform | Week 10.
  Number of characters submitted in the internet treatment platform. Separate data for children and parents.
The Child and Adolescent Gilles de la Tourette Syndrome-Quality of Life Scale (C&A-GTS-QOL) | Baseline; week 10; 3-month follow-up; 6-month follow-up; 12-month follow-up.
  Used to assess disease-specific health-related quality of life. Two different versions will be used, one for participants aged 9-12, and one for participants aged 13-17. Child/adolescent-reported.
Short Mood and Feeling Questionnaire - child version (SMFQ) + additional suicide item | Baseline; mid-treatment (5 weeks post-baseline); week 10; 3-month follow-up; 6-month follow-up; 12-month follow-up.
  Used to assess depressive symptoms and suicidal ideation. Child/adolescent-reported.
Obsessive-compulsive inventory - child version (OCI-CV) | Baseline; week 10; 3-month follow-up; 6-month follow-up; 12-month follow-up.
  Used to assess obsessive-compulsive symptoms. Child/adolescent-reported.
Treatment credibility questionnaire | Mid-treatment (3 weeks post-baseline).
  Questionnaire developed by the research team. Used to assess treatment credibility. Separate versions for the child/adolescent and the parent are used.
Working alliance inventory - child and parent versions (WAI-C and WAI-P ) | Mid-treatment (3 weeks post-baseline).
  Used to assess the child/adolescent/parent's perceived working alliance with their therapist. Separate versions for the child/adolescent and the parent are used.
Treatment satisfaction questionnaire | 3-month follow-up.
  Questionnaire developed by the research team. Used to assess treatment satisfaction. Separate versions for the child/adolescent and the parent are used.
KIDSCREEN-10 | Baseline; week 10; 3-month follow-up; 6-month follow-up; 12-month follow-up.
  Used to assess quality of life, with the intention to transform this data into quality adjusted lifetime years (QALYs). Separate versions for the child/adolescent and the parent are used.
Parent Tic Questionnaire (PTQ) | Baseline; mid-treatment (5 weeks post-baseline); week 10; 3-month follow-up; 6-month follow-up; 12-month follow-up.
  Used to assess tic severity. Parent-reported.
Short Mood and Feeling Questionnaire - parent version (SMFQ) | Baseline; mid-treatment (5 weeks post-baseline); week 10; 3-month follow-up; 6-month follow-up; 12-month follow-up.
  Used to assess depressive symptoms. Parent-reported.
Side effects questionnaire | Baseline; mid-treatment (5 weeks post-baseline); week 10; 3-month follow-up.
  Used to assess side effects/adverse events for the child/adolescent. Parent-reported.
Trimbos Questionnaire for Costs associated with Psychiatric Illness (TiC-P) | Baseline; week 10; 3-month follow-up; 6-month follow-up; 12-month follow-up.
  Used to assess healthcare and societal resource use. Parent-reported.

CONTACTS AND LOCATIONS:
Overall Officials: David Mataix-Cols, PhD, Principal Investigator — Department of Clinical Neuroscience (CNS), Karolinska Institutet
Locations (1):
- Child and Adolescent Psychiatry Research Center, BUP Klinisk forskningsenhet, Stockholm, Sweden

REFERENCES:
- [Background] Andren P, Aspvall K, Fernandez de la Cruz L, Wiktor P, Romano S, Andersson E, Murphy T, Isomura K, Serlachius E, Mataix-Cols D. Therapist-guided and parent-guided internet-delivered behaviour therapy for paediatric Tourette's disorder: a pilot randomised controlled trial with long-term follow-up. BMJ Open. 2019 Feb 15;9(2):e024685. doi: 10.1136/bmjopen-2018-024685. PMID 30772854
- [Derived] Andren P, Sampaio F, Ringberg H, Wachtmeister V, Warnstrom M, Isomura K, Aspvall K, Lenhard F, Hall CL, Davies EB, Murphy T, Hollis C, Feldman I, Bottai M, Serlachius E, Andersson E, Fernandez de la Cruz L, Mataix-Cols D. Internet-Delivered Exposure and Response Prevention for Pediatric Tourette Syndrome: 12-Month Follow-Up of a Randomized Clinical Trial. JAMA Netw Open. 2024 May 1;7(5):e248468. doi: 10.1001/jamanetworkopen.2024.8468. PMID 38700867
- [Derived] Andren P, Holmsved M, Ringberg H, Wachtmeister V, Isomura K, Aspvall K, Lenhard F, Hall CL, Davies EB, Murphy T, Hollis C, Sampaio F, Feldman I, Bottai M, Serlachius E, Andersson E, Fernandez de la Cruz L, Mataix-Cols D. Therapist-Supported Internet-Delivered Exposure and Response Prevention for Children and Adolescents With Tourette Syndrome: A Randomized Clinical Trial. JAMA Netw Open. 2022 Aug 1;5(8):e2225614. doi: 10.1001/jamanetworkopen.2022.25614. PMID 35969401
- [Derived] Andren P, Fernandez de la Cruz L, Isomura K, Lenhard F, Hall CL, Davies EB, Murphy T, Hollis C, Sampaio F, Feldman I, Bottai M, Serlachius E, Andersson E, Mataix-Cols D. Efficacy and cost-effectiveness of therapist-guided internet-delivered behaviour therapy for children and adolescents with Tourette syndrome: study protocol for a single-blind randomised controlled trial. Trials. 2021 Sep 30;22(1):669. doi: 10.1186/s13063-021-05592-z. PMID 34593015